CLINICAL TRIAL: NCT02851641
Title: Risk and Importance of Peroperative Nasal Hemorrhage in the Treatment of Lacrimal Duct Obstruction in Young Children
Acronym: CANALHEMO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CEN_2015_9
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Lacrimal Duct Obstruction
MeSH Terms: conditions — Lacrimal Duct Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Nasolacrimal duct obstruction
  Interventions: Procedure: "pushed" mono-canaliculonasal intubation

INTERVENTIONS:
Procedure: "pushed" mono-canaliculonasal intubation

SUMMARY:
The aim of the study is to evaluate the risk in intra-operative nasal hemorrhage when using a "pushed" probe (Master Ka) in the treatment of naso lacrimal duct obstruction (NLDO).

In the investigator's experience, this risk seemed to minus using a pushed probe rather than the classical pulled-type probes.

A lower risk of hemorrhage could lead to a change in the anesthetic procedure. The gold standard in NLDO is the use of an orotracheal intubation. It could then be replaced by the use of an orolaryngeal mask. A forthcoming study will evaluate the results of this anesthetic change.

ELIGIBILITY:
Inclusion Criteria:

* < 6 years of age
* Unilateral lacrimal duct obstruction with programmed surgery
* Surgery scheduled wih a "pushed" mono-canaliculonasal intubation
* No opposition of parents for he participation of their child

Exclusion Criteria:

* Coagulation disorder
* Previous history of nasolacrimal intubation (homo or contra-lateral)
* Non covered by health insurance

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with congenital nasolacrimal duct obstruction
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Nasal hemorrhage | Through surgery completion, an average of 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France